CLINICAL TRIAL: NCT06765031
Title: The Role of Furosemide Stress Test in Predicting Acute Kidney Injury Progression and Need for Renal Replacement Therapy in Patients Followed in the Intensive Care Clinic
Brief Title: The Role of Furosemide Stress Test in the Intensive Care Clinic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Mete Erdemir, principal investigator, Gulhane Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: AEŞH-BADEK-2024-1037
Record Dates: First submitted 2024-12-19; First posted 2025-01-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Akut Kidney Injury
Keywords: akut kidney injury; furosemide stres test; continuous renal replasman terapy
MeSH Terms: interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Furosemide stress test application in AKI stage 1-2 according to kdigo criteria (Other): Among the patients included in the study, furosemide will be administered intravenously as a push at a dose of 1 mg/kg to patients who have not used furosemide in the last 7 days within the first 24 hours following ICU admission, and at a dose of 1.5 mg/kg to patients who have been exposed to furosemide. Patients who can pass 200 ml or more of urine within the first 2 hours after furosemide administration will be evaluated as having a positive furosemide stress test.
  Interventions: Drug: Furosemide

INTERVENTIONS:
Drug: Furosemide — Furosemide will be administered intravenously in the form of a push at a dose of 1 mg/kg to furosemide-naïve patients who meet the inclusion criteria and at a dose of 1.5 mg/kg to patients exposed to furosemide.

SUMMARY:
AKI causes high mortality and morbidity, especially in critically ill patients, and prolongs the patient's stay in the intensive care unit. Due to the high morbidity and mortality associated with AKI, many researchers are studying several new biomarkers for earlier detection of AKI, determination of etiologies, and prediction of outcomes. However, the use of these new biomarkers may be limited due to reimbursement issues. In addition to the therapeutic role of furosemide in fluid balance, blood pressure control, and hypercalcemia management, Chawla et al. recommend the furosemide stress test (FST) as a tool to predict AKI progression. Designing a test that predicts the probability of AKI progression will help us make better decisions regarding the optimal timing of RRT initiation. In this study, we aimed to evaluate the feasibility of using the FST test in determining the progression of AKI in patients hospitalized in the intensive care unit and the need for RRT using the noninvasive procedure furosemide stress test.

DETAILED DESCRIPTION:
Acute kidney injury is defined by the KDIGO guidelines as an increase in serum creatinine ≥0.3 mg/dL (≥26.5 μmol/L) within the previous 48 hours, a ≥1.5-fold increase in serum creatinine from baseline that is known or presumed to have occurred within the previous seven days, or a urine volume of <0.5 mL/kg/h over six hours. In addition to the therapeutic role of furosemide in fluid balance, blood pressure control, and management of hypercalcemia, Chawla et al. recommend the furosemide stress test (FST) as a tool to predict AKI progression . Patients who develop AKI often require renal replacement therapy (RRT), but there is often no consensus on the optimal timing of initiation of RRT. RRT is an invasive procedure. The goal in AKI patients is to restore kidney function to normal without invasive intervention. However, a more conservative approach to starting RRT during the course of AKI may expose the patient to adverse outcomes. Therefore, designing a test that predicts the possibility of more severe AKI progression will help us make better decisions about the optimal timing of starting RRT. Albumin, sodium, potassium, chloride, magnesium, creatinine, glomerular filtration rate, urea and venous blood gases will be studied from the residual blood of the patients before FST. Creatinine, sodium, potassium, urea and microalbumin levels will be studied in the spot urine of the patients from the residual urine before FST. Fractional sodium-urea levels will be calculated with these results. The total urine volume will be calculated by collecting the 1st and 2st hour urines separately after FST and also the Na concentration will be measured from these urine samples. Systolic, diastolic and mean blood pressure levels obtained from the right arm with a noninvasive method (with a cuff) at the time of FST will be noted. In addition, persistent AKI risk index (PERSANT AKI risk index (PARI)), eGFR and kinetic GFR will be calculated and noted simultaneously with FST. Demographic data of the patients will be obtained from the hospital system. The lowest creatinine level in the last 6 months before application of the patients accepted to the study will be accepted as the basal creatinine level. If the creatinine level taken in the last 6 months cannot be reached, the lowest creatinine level reached before application will be accepted as the basal creatinine level.

Among the patients included in the study, 1 mg/kg furosemide will be administered to patients who have not used furosemide in the last 7 days within the first 24 hours following ICU admission, and 1.5 mg/kg furosemide will be administered intravenously as a push in patients exposed to furosemide. Patients who can pass 200 ml or more urine within the first 2 hours after furosemide application will be evaluated as positive for furosemide stress test.

Progression from AKI stage 1-2 to AKI stage 3 within 14 days after FST, need for RRT, total intensive care unit stay, development of persistent acute kidney injury (PAKi), number of RRT-independent days, renal recovery time and all-cause mortality will be evaluated

ELIGIBILITY:
Inclusion Criteria:

1. Those who meet KDIGO AKI stage 1 and stage 2 criteria in the first 24 hours
2. Those with sufficient fluid volume (CVP≥6 cmH20)
3. Female and male patients over the age of 18 will be included in the study

Exclusion Criteria:

1. Pregnant patients
2. Hospitalization due to intoxication
3. Liver or kidney transplant
4. Glomerular filtration rate below 30 ml/min/1.73m2
5. Active bleeding
6. Patients with obstructive uropathy
7. Patients in need of urgent RRT (K≥6.6 meq/L, pH<7.15, pulmonary edema due to fluid overload, uremic complications)
8. Patients evaluated as KDIGO AKI stage 3
9. Patients who have received RRT in the last 30 days
10. Patients with CKD diagnosis
11. Patients with pulmonary embolism
12. Hypoalbuminemia≥2.5 g/dl,
13. Patients receiving cephalosporin treatment will be excluded from the sample.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Progression from AKI Stage 1-2 to Stage 3 within 14 days in patients who underwent furosemide stress test | 14 days after FST
  Among the patients included in the study, within the first 24 hours following ICU admission, patients who have not used Furosemide within the last 7 days will be administered 1 mg/kg intravenously as a push for patients who have been exposed to furosemide, and 1.5 mg/kg for patients who have been exposed to furosemide. Patients who can excrete 200 ml or more urine within the first 2 hours after furosemide administration will be evaluated as having a positive furosemide stress test(FST). Our primary outcome is to determine how helpful it is in predicting progression from AKI stage 1-2 to AKI stage 3 within 14 days after the FST.

SECONDARY OUTCOMES:
Renal Replacement Therapy | Within 14 days post-FST
  Incidence of patients requiring initiation of CRRT based on clinical indications
Persistent AKI | Up to 14 days post-FST
  Proportion of patients whose AKI persists beyond 48 hours from the Furosemide Stress Test, as defined by KDIGO criteria.
Hospital Stay | From date of FST until discharge or death (up to 90 days)
  Total number of days spent in the hospital following the Furosemide Stress Test.
Mortality | 28 days post-FST
  All-cause mortality rate recorded within 28 days after the FST.

CONTACTS AND LOCATIONS:
Overall Officials: gürhan t taşkın, Associate Professor, Study Director — Gulhane Training and Research Hospital
Locations (1):
- Gulhane Training and Research Hospital, Ankara, keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Result] Chawla LS, Davison DL, Brasha-Mitchell E, Koyner JL, Arthur JM, Shaw AD, Tumlin JA, Trevino SA, Kimmel PL, Seneff MG. Development and standardization of a furosemide stress test to predict the severity of acute kidney injury. Crit Care. 2013 Sep 20;17(5):R207. doi: 10.1186/cc13015. PMID 24053972
- [Result] Gibney N, Hoste E, Burdmann EA, Bunchman T, Kher V, Viswanathan R, Mehta RL, Ronco C. Timing of initiation and discontinuation of renal replacement therapy in AKI: unanswered key questions. Clin J Am Soc Nephrol. 2008 May;3(3):876-80. doi: 10.2215/CJN.04871107. Epub 2008 Mar 5. PMID 18322044